CLINICAL TRIAL: NCT01997359
Title: Multi-level Determinants of Starting ART Late in Sub-Saharan Africa (LSTART Study): A Case-control Study to Identify Individual-level Risk Factors for Late ART Initiation in Ethiopia
Brief Title: Multi-level Determinants of Starting ART Late: Aim 3
Acronym: LSTART
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Batya Elul, Assistant Professor of Clinical Epidemiology, Columbia University
Other Study IDs: AAAI1960; 1R01MH089831 (NIH)
Record Dates: First submitted 2013-11-08; First posted 2013-11-28 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Human Immunodeficiency Virus (HIV); Acquired Immune Deficiency Syndrome (AIDS)
Keywords: ART initiation; HIV; AIDS; Ethiopia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Key Informant Interviews: Eligible patients will undergo a one hour structured interview about barriers and facilitators to early ART initiation.
- Prospective Cohort: The prospective cohort will include all patients initiating ART at one of the six study sites, estimated at 1,200 patients. Cases will be adults initiating ART with either: CD4 count <150 cells/µL. Controls will be adults who initiate ART with CD4≥200 . Individuals initiating ART with CD4 counts of 150-199 cells per µL and at WHO Stage I-III will be excluded from the case-control analysis in order to ensure meaningful distinction between the two groups. We will enroll 720 patients for the case control study nested in the prospective cohort, which will include 360 cases and 360 controls, who will be frequency matched by sex, month of ART initiation, and clinic.

SUMMARY:
The availability of HIV care and treatment programs is increasing in sub-Saharan Africa. However more than half the patients who need HIV treatment are still not receiving antiretroviral therapy (ART). This can lead to early death from AIDS. Additionally, many patients start ART late after the HIV disease is very advanced. This results in high death rates soon after starting ART. The factors that contribute to late ART initiation are still unclear. This study will identify factors that help patients to enroll or prevent them from enrolling into HIV care and starting ART on time. We will examine the characteristics of all patients initiating ART at study sites. We will also look at potential risk factors among patients who initiate ART late (cases) compared to patients who initiate earlier (controls) at 6 HIV care and treatment clinics in Ethiopia. Data will be collected using 2 methods:

1. Face-to-face interviews with participants using questionnaires
2. Obtaining clinical data from the electronic patient-level database

Identifying factors that help patients to start or prevent them from starting ART on time will help to direct interventions, programs and policies to reduce early death.

DETAILED DESCRIPTION:
Background: Although HIV care and treatment programs are being scaled up in sub-Saharan Africa, more than 50% of the patients in need of ART are not receiving it and there is still significant mortality from AIDS. One of the major challenges is high rates of late ART initiation (i.e., in the advanced stages of HIV disease) which results in high rates of mortality soon after initiation of ART. The individual-level factors that contribute to late ART initiation are still unclear. Objective: As the 3rd part of a 3-phase NIH-sponsored project, this study aims to identify individual-level enablers and barriers to timely enrollment into HIV care and ART initiation.

Methods: We will be recruiting all patients newly initiating ART at the study sites for descriptive analysis (approximately 1,200). As a sub-analysis, we will be utilizing a case-control approach to examine potential individual risk factors (e.g. knowledge and behaviors around HIV care and treatment, experience of stigma, and other perceived barriers and enablers to earlier HIV diagnosis, enrollment into care, and ART initiation) among 360 patients who initiated ART late (CD4 count <150 cells/µL compared to 360 patients who initiated earlier (CD4≥200) at 6 HIV care and treatment clinics in Ethiopia. For both the descriptive study and case-control study, data will be collected using 2 methods:

1. Face-to-face interviews with participants using structured questionnaires
2. Abstraction of clinical data from the electronic patient-level database to capture patient information at baseline, 6 and 12 months after enrollment in the study

Expected use of results: Identifying individual-level enablers and barriers of timely ART initiation will facilitate implementation of interventions, programs and policies to mitigate the problem of late ART initiation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years (the age of majority in Ethiopia) or older.
* ART naïve.
* Eligible for ART according to Ethiopia's National ART guideline criteria.
* Have received a prescription for ART during the study period.
* Speak either Oromiffa or Amharic.
* Special inclusion criteria for case-control sub-analysis:

  * Cases: CD4 count <150 cells/µL (regardless of WHO stage)
  * Controls: CD4 ≥200.

Exclusion Criteria:

* Overtly cognitively impaired
* Inability or unwillingness to provide informed consent
* Actively incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective cohort will include all patients initiating ART at one of the six study sites, estimated at 1,200 patients. Cases will be adults initiating ART with either: CD4 count <150 cells/µL. Controls will be adults who initiate ART with CD4≥200 . Individuals initiating ART with CD4 counts of 150-199 cells per µL and at WHO Stage I-III will be excluded from the case-control analysis in order to ensure meaningful distinction between the two groups. We will enroll 720 patients for the case control study nested in the prospective cohort, which will include 360 cases and 360 controls, who will be frequency matched by sex, month of ART initiation, and clinic.
Sampling Method: Non-Probability Sample
Enrollment: 1214 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of Persons Initiating ART Late | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Batya Elul, PhD, MSc, Principal Investigator — ICAP-NY, Columbia University
Locations (6):
- Ethiopia (6):
  - Ambo Hospital, Āmbo
  - Bishoftu Hospital, Bishoftu
  - Fitche Hospital, Fichē
  - Goba Hospital, Goba
  - Nekemte Hospital, Nekemte
  - Shashamene Hospital, Shashamene